CLINICAL TRIAL: NCT00211887
Title: A Multi-Center, Double-Blind, Randomized Study Comparing the Combined Use of Interferon Beta-1a and Glatiramer Acetate to Either Agent Alone in Patients With Relapsing-Remitting Multiple Sclerosis (CombiRx)
Brief Title: Combination Therapy in Patients With Relapsing-Remitting Multiple Sclerosis (MS)CombiRx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Lublin (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Fred Lublin, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 02-0526; 02-0526; CRC; U01NS045719 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Clinical trial; treatment trial; autoimmune disease; Relapsing Remitting; MS Treatment; interferon beta-1a; glatiramer acetate
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Autoimmune Diseases | interventions — Interferon beta-1a; Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interferon beta 1-a (Active Comparator): Active Interferon B1a Weekly vs. Placebo Glatiramer Acetate
  Interferon b-1a (IFN) intramuscularly weekly
  Interventions: Drug: Interferon beta 1-a; Other: placebo
- glatiramer acetate (Active Comparator): Placebo Interferon B1a Weekly vs. Active Glatiramer Acetate
  Glatiramer acetate 20mg daily
  Interventions: Drug: glatiramer acetate; Other: placebo
- IFN and GA (Active Comparator): Active Interferon B1a Weekly and Active Glatiramer Acetate
  Interventions: Drug: Interferon beta 1-a; Drug: glatiramer acetate

INTERVENTIONS:
Drug: Interferon beta 1-a — The single agent arm is divided into two groups, IFN and GA providing for 3 treatment arms: IFN IM and GA SC (50% of the patients), IFN IM and placebo SC (25% of the patients) and GA SC and placebo IM (25% of the patients).
  Other Names: IFN
  Arms: IFN and GA; Interferon beta 1-a
Drug: glatiramer acetate — The single agent arm is divided into two groups, IFN and GA providing for 3 treatment arms: IFN IM and GA SC (50% of the patients), IFN IM and placebo SC (25% of the patients) and GA SC and placebo IM (25% of the patients).
  Other Names: GA
  Arms: IFN and GA; glatiramer acetate
Other: placebo — an inactive substance
  Arms: Interferon beta 1-a; glatiramer acetate

SUMMARY:
This is for a randomized clinical trial (RCT) to determine if the combined use of interferon beta-1a (IFN) and glatiramer acetate (GA) is a measurably better therapy than either agent used individually in patients with relapsing-remitting (RR) multiple sclerosis (MS).

DETAILED DESCRIPTION:
This is a multicenter, double blind, randomized trial examining combination therapy versus single agent therapy with three-year follow-up on the last patient randomized. All patients will remain on therapy until the last patient completes the study. All patients will then be transitioned, based on the findings, to open label of combination with continued follow-up or some recommendation about single agent therapy. While the study design benefits from having two arms of single agent therapy to examine the important question of whether there are differences between the single agents, the primary interest is in combination therapy. Therefore, a two-group combination versus single agent concept was used - splitting the population into single agent and combination therapy equally. The single agent arm is divided into two groups, IFN and GA providing for 3 treatment arms: IFN intramuscularly (IM) and GA subcutaneously (SC) (50% of the patients), IFN IM and placebo SC (25% of the patients) and GA SC and placebo IM (25% of the patients).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 and 60 years, inclusive.
* Diagnosis of relapsing-remitting MS by either the Poser or McDonald criteria.
* Expanded Disability Status Scale (EDSS) score between 0 and 5.5, inclusive.
* At least 2 exacerbations in the prior three years; one exacerbation may utilize the McDonald MRI criteria for dissemination in time (a new gadolinium [Gd]-enhancing lesion demonstrated on a scan done at least 3 months following onset of a clinical attack or a new T2 lesion or Gd-enhancing lesion on a follow-up scan after an additional 3 months).
* Give written informed consent prior to any testing under this protocol, including screening tests and evaluations that are not considered part of the subject's routine care.

Exclusion Criteria:

* Any prior use of interferon beta or glatiramer acetate.
* Acute exacerbation within 30 days of screening.
* Steroids for acute exacerbations (>100 mg/day) within 30 days of study entrance or chronic systemic steroid use.
* Evidence of progressive MS.
* Use IVIg, azathioprine, methotrexate, cyclosporine, mitoxantrone, cyclophosphamide, mycophenolate (CellCept) or plasma exchange in the twelve weeks prior to study drug dosing.
* Any previous treatment with natalizumab (Tysabri, Antegren), cladribine, T cell vaccine, Campath, daclizumab, rituximab, altered peptide ligand or total lymphoid irradiation.
* Treatment with 4 aminopyridines in the four weeks prior to study drug dosing.
* Prior treatment with any other investigational drug, unless approved by the Clinical Coordinating Center (Dr. Lublin).
* Inability to perform the baseline MSFC (timed 25-foot walk, 9-hole peg test [9HPT], and Paced Auditory Serial Addition Test 3 [PASAT3]).
* Inability to undergo baseline MRI scan.
* History of any significant cardiac, hepatic, pulmonary, or renal disease, immune deficiency, or other medical conditions that would preclude therapy with interferon beta, glatiramer acetate, or participation in this study.
* Known history of sensitivity to gadopentetate dimeglumine or mannitol.
* History of a seizure within the 3 months prior to randomization.
* History of suicidal ideation or an episode of severe depression within the 3 months prior to randomization.
* Abnormal screening blood tests exceeding any of the limits defined below:

  * Alanine transaminase (ALT) or aspartate transaminase (AST) greater than two times the upper limit of normal (i.e., >2 × ULN)
  * Total white blood cell count <2,300/mm3
  * Platelet count <80,000/mm3
  * Creatinine >2 × ULN
* Participation in another experimental clinical trial, without formal approval.
* History of alcohol or drug abuse within the 2 years prior to randomization.
* Female subjects who are currently pregnant, breast-feeding, or plan to become pregnant.
* For female subjects, unless postmenopausal or surgically sterile, unwillingness to practice effective contraception, as defined by the investigator, during the study. The rhythm method is not to be used as the sole method of contraception.
* Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition that is likely to affect the subject's returning for scheduled follow-up visits on schedule (any physical, mental, or social condition).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1008 (Actual)
Dates: Start 2005-01; Primary Completion 2012-04 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Lublin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (71):
- United States (67):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Barrow Neurology Clinic, Phoenix, Arizona
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - Northwest Neurospecialists PLLC, Tucson, Arizona
  - Sutter East Bay Medical Group, Berkeley, California
  - Neurology Center North Orange County, La Habra, California
  - VA West Los Angeles Healthcare Center, Los Angeles, California
  - University of California - Davis Medical Center, Sacramento, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Patricia Fodor P.C., Colorado Springs, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Neurology Associates, PA, Maitland, Florida
  - University of Miami - Neurology, Miami, Florida
  - MS Center of Atlanta, Atlanta, Georgia
  - Shepherd Center, Atlanta, Georgia
  - Northwest University, Chicago, Illinois
  - Consultants in Neurology - Multiple Sclerosis Center, Northbrook, Illinois
  - University of Illinois College of Medicine, Peoria, Illinois
  - Ruan Neurology Clinic and Research Center, Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Maryland Center for MS, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Minneapolis Clinic - MS Center, Golden Valley, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - St. Louis University - St. Louis VA, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Northern Rockies MS Center, Billings, Montana
  - Dartmouth Medical School, Lebanon, New Hampshire
  - CentraState Medical Center, Freehold, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Neuro Associates of Albany, PC, Albany, New York
  - Albany Medical College, Albany, New York
  - The Jacobs Neurological Institute, Buffalo, New York
  - Winthrop Neurology Faculty Practice, Mineola, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - NYU Hospital For Joint Diseases, New York, New York
  - South Shore Neurologic Associates Inc., Patchogue, New York
  - University of Rochester, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - CMC-Neuroscience & Spine Institute, Division of Neurology, MS Center, Charlotte, North Carolina
  - Meritcare Neuroscience, Fargo, North Dakota
  - NeuroCare Center, Inc., Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Neurology Specialists, Dayton, Ohio
  - Medical College Of Ohio, Toledo, Ohio
  - Oak Clinic for Multiple Sclerosis, Uniontown, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny MS Treatment Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Neurological Research Center, Inc., Bennington, Vermont
  - Fletcher Allen Health Care, Burlington, Vermont
  - Neurological Associates, Inc., Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - MS Center at Evergreen, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
  - Regional MS Center at St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - Capital Health and the University of Alberta, Edmonton, Alberta
  - Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital-Multiple Sclerosis Research Center, Toronto, Ontario

REFERENCES:
- [Result] Lublin FD, Cofield SS, Cutter GR, Conwit R, Narayana PA, Nelson F, Salter AR, Gustafson T, Wolinsky JS; CombiRx Investigators. Randomized study combining interferon and glatiramer acetate in multiple sclerosis. Ann Neurol. 2013 Mar;73(3):327-40. doi: 10.1002/ana.23863. Epub 2013 Mar 11. PMID 23424159
- [Derived] Koch MW, Moral E, Brieva L, Mostert J, Strijbis EM, Comtois J, Repovic P, Bowen JD, Wolinsky JS, Lublin FD, Cutter G. Relapse recovery in relapsing-remitting multiple sclerosis: An analysis of the CombiRx dataset. Mult Scler. 2023 Dec;29(14):1776-1785. doi: 10.1177/13524585231202320. Epub 2023 Oct 13. PMID 37830451
- [Derived] Satyanarayan S, Cutter G, Krieger S, Cofield S, Wolinsky JS, Lublin F. The impact of relapse definition and measures of durability on MS clinical trial outcomes. Mult Scler. 2023 Apr;29(4-5):568-575. doi: 10.1177/13524585231157211. PMID 37119208
- [Derived] Zhang Y, Cofield S, Cutter G, Krieger S, Wolinsky JS, Lublin F. Predictors of Disease Activity and Worsening in Relapsing-Remitting Multiple Sclerosis. Neurol Clin Pract. 2022 Aug;12(4):e58-e65. doi: 10.1212/CPJ.0000000000001177. PMID 36382118
- [Derived] Koch MW, Mostert J, Repovic P, Bowen JD, Wolinsky JS, Lublin FD, Strijbis E, Cutter G. Early first-line treatment response and subsequent disability worsening in relapsing-remitting multiple sclerosis. Eur J Neurol. 2022 Apr;29(4):1106-1116. doi: 10.1111/ene.15220. Epub 2021 Dec 26. PMID 34927308
- [Derived] Ben-Zacharia AB, Janal MN, Brody AA, Wolinsky J, Lublin F, Cutter G. The Effect of Body Mass Index on Brain Volume and Cognitive Function in Relapsing-Remitting Multiple sclerosis: A CombiRx Secondary Analysis. J Cent Nerv Syst Dis. 2021 Nov 6;13:11795735211042173. doi: 10.1177/11795735211042173. eCollection 2021. PMID 34759712
- [Derived] Petracca M, Cutter G, Cocozza S, Freeman L, Kangarlu J, Margoni M, Moro M, Krieger S, El Mendili MM, Droby A, Wolinsky JS, Lublin F, Inglese M. Cerebellar pathology and disability worsening in relapsing-remitting multiple sclerosis: A retrospective analysis from the CombiRx trial. Eur J Neurol. 2022 Feb;29(2):515-521. doi: 10.1111/ene.15157. Epub 2021 Nov 17. PMID 34695274
- [Derived] Koch MW, Mostert JP, Wolinsky JS, Lublin FD, Uitdehaag B, Cutter GR. Comparison of the EDSS, Timed 25-Foot Walk, and the 9-Hole Peg Test as Clinical Trial Outcomes in Relapsing-Remitting Multiple Sclerosis. Neurology. 2021 Oct 19;97(16):e1560-e1570. doi: 10.1212/WNL.0000000000012690. Epub 2021 Aug 25. PMID 34433679
- [Derived] Koch MW, Mostert J, Zhang Y, Wolinsky JS, Lublin FD, Strijbis E, Cutter G. Association of Age With Contrast-Enhancing Lesions Across the Multiple Sclerosis Disease Spectrum. Neurology. 2021 Sep 28;97(13):e1334-e1342. doi: 10.1212/WNL.0000000000012603. Epub 2021 Aug 10. PMID 34376508
- [Derived] Salter A, Kowalec K, Fitzgerald KC, Cutter G, Marrie RA. Comorbidity is associated with disease activity in MS: Findings from the CombiRx trial. Neurology. 2020 Aug 4;95(5):e446-e456. doi: 10.1212/WNL.0000000000010024. Epub 2020 Jun 17. PMID 32554770
- [Derived] Fitzgerald KC, Kim K, Smith MD, Aston SA, Fioravante N, Rothman AM, Krieger S, Cofield SS, Kimbrough DJ, Bhargava P, Saidha S, Whartenby KA, Green AJ, Mowry EM, Cutter GR, Lublin FD, Baranzini SE, De Jager PL, Calabresi PA. Early complement genes are associated with visual system degeneration in multiple sclerosis. Brain. 2019 Sep 1;142(9):2722-2736. doi: 10.1093/brain/awz188. PMID 31289819
- [Derived] Bhanushali MJ, Gustafson T, Powell S, Conwit RA, Wolinsky JS, Cutter GR, Lublin FD, Cofield SS. Recruitment of participants to a multiple sclerosis trial: the CombiRx experience. Clin Trials. 2014 Apr;11(2):159-66. doi: 10.1177/1740774513517184. PMID 24686106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial enrolled participants from January 2005 through April 2009. The trial was conducted in 68 sites, both private practice and academic, in the USA and Canada.
Pre-assignment Details: 1129 participants assessed for eligibility. 121 excluded due to recent activity (16), <2 exacerbations (14), other medical exclusions (14), inconclusive for RRMS (12), abnormal lab value (10), cannot have Gd (5), EDSS>5.5 (2), and other reason (46).
Groups:
- IFN + GA: Interferon beta-1a 30µg intramuscularly weekly and glatiramer acetate (GA) 20mg daily
- Interferon Beta 1a: Interferon beta-1a 30µg intramuscularly weekly
- Glatiramer Acetate: glatiramer acetate 20mg daily
Period: Overall Study
Arm/Group | IFN + GA | Interferon Beta 1a | Glatiramer Acetate
Started | 499 | 250 | 259
Completed | 397 | 194 | 223
Not Completed | 102 | 56 | 36
Not completed — Adverse Event | 8 | 4 | 6
Not completed — Death | 1 | 1 | 1
Not completed — Lost to Follow-up | 28 | 13 | 9
Not completed — Non-medical reason | 31 | 14 | 8
Not completed — Other medical reason | 15 | 11 | 7
Not completed — Side effects | 19 | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- IFN + GA: Interferon beta-1a intramuscularly weekly and glatiramer acetate daily
- IFB-1a: Interferon beta-1a
- Glatiramer: glatiramer acetate
- Total: Total of all reporting groups
Arm/Group | IFN + GA | IFB-1a | Glatiramer | Total
Number analyzed (Participants) | 499 | 250 | 259 | 1008
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (9.4) | 37.6 (10.2) | 39.0 (9.5) | 37.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 372 | 173 | 185 | 730
  Male | 127 | 77 | 74 | 278

OUTCOME MEASURES:

1. Primary Outcome: ARR - PDEs
Description: Annualized relapse rate of protocol-defined exacerbations Protocol defined relapse - an relapse seen within 7 days of onset, verified by the treating physician and independently observed as a change in EDSS by the examining physician. This relapse is defined as: the appearance of a new symptom or worsening of an old symptom, attributable to MS; accompanied by a change in the neurologic examination (defined as a 0.5 or greater increase in the EDSS over the last scheduled or unscheduled visit or a 2 point change in one functional system or a 1 point change in two functional systems, except bladder and cognitive changes); lasting at least 24 hours in the absence of fever; and preceded by stability or improvement for at least 30 days.
Time Frame: Baseline to Month 36
Measure: Number; unit: relapses per year
Arm/Group | IFN + GA | IFB-1a | Glatiramer
Number analyzed (Participants) | 499 | 250 | 259
relapses per year | 0.12 | 0.16 | 0.11

2. Secondary Outcome: Confirmed Progression on the Expanded Disability Status Scale
Description: % with EDSS progression
  Confirmed progression in a participant was defined as a 1.0 increase in the EDSS from baseline, when baseline <=5.0; or an increase of 0.5 from baseline, when baseline >=5.5, sustained for 6 months (2 successive quarterly visits), as assessed by the blinded EDSS examiner and confirmed centrally.
Time Frame: Baseline to Month 36
Measure: Number; unit: percentage of participants
Arm/Group | IFN + GA | IFB-1a | Glatiramer
Number analyzed (Participants) | 499 | 250 | 259
percentage of participants | 23.9 (1.2) | 21.6 (1.2) | 24.8 (1.2)

3. Secondary Outcome: Change in the Multiple Sclerosis Functional Composite
Description: positive indicates improvement
  The Multiple Sclerosis Functional Composite (MSFC) is a scale measuring pyramidal functions, sensory functions, cerebellar functions, bowel & bladder functions,brain stem functions, mental functions, and visual functions from 0 to 6.
  0= normal 6= severe loss
Time Frame: Baseline to month 36
Population: Due to participant dropouts, there were less participants analyzed for this particular outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IFN + GA | IFB-1a | Glatiramer
Number analyzed (Participants) | 472 | 241 | 246
units on a scale | 0.1 (0.5) [-3.5 to 2.3] | 0.1 (0.5) [-2.0 to 1.8] | 0.2 (0.5) [-3.0 to 2.4]

4. Secondary Outcome: Change in MRI Composite Score
Description: MRI composite score (Z4 score) - the unweighted sum of the individual Z scores for enhanced tissue volume, T2 lesion burden, equivalence of the T1 hypointense lesion burden, normalized CSF (an inverse measure of atrophy with the appropriate sign so that all scores are directionally compatible - larger is worse) MRI enhancement status at baseline (0, 1-4, and 5 or more enhancing lesions)
Time Frame: Baseline to month 36
Population: Due to participant dropouts, there were less participants analyzed for this particular outcome measure.
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | IFN + GA | IFB-1a | Glatiramer
Number analyzed (Participants) | 381 | 185 | 211
z score | -0.02 (1.30) | 0.05 (1.27) | 0.10 (2.09)

ADVERSE EVENTS:
Description: Adverse events were only collected with regard to the affected organ system.
Arm/Group | IFN + GA | IFB-1a | Glatiramer
Serious Adverse Events (participants affected / at risk) | 70/499 | 38/250 | 30/259
Other Adverse Events (participants affected / at risk) | 197/499 | 102/250 | 98/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFN + GA (N=499) | IFB-1a (N=250) | Glatiramer (N=259)
Cardiac disorders (Cardiac disorders) | 3 (3) | 3 (3) | 3 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 7 (7) | 3 (3) | 2 (2)
Hepato-biliary disorders (Hepatobiliary disorders) | 4 (4) | 1 (1) | 3 (3)
Infections and infestations (Infections and infestations) | 11 (11) | 4 (4) | 1 (1)
Musculoskeletal, connective tissue and bone disorders (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (2)
Neoplasms benign and malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6) | 3 (3)
Nervous system disorders (Nervous system disorders) | 17 (17) | 11 (11) | 5 (5)
Psychiatric disorders (Psychiatric disorders) | 15 (15) | 4 (4) | 8 (8)
Renal and urinary disorders (Renal and urinary disorders) | 3 (3) | 3 (3) | 0 (0)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 3 (3) | 2 (2) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 9 (9) | 5 (5) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFN + GA (N=499) | IFB-1a (N=250) | Glatiramer (N=259)
constipation (Gastrointestinal disorders) | 23 (29) | 19 (20) | 18 (19)
Diarrhea (Gastrointestinal disorders) | 32 (36) | 21 (27) | 20 (20)
GI Upset (Gastrointestinal disorders) | 41 (44) | 11 (12) | 13 (15)
Nausea/Vomiting (Gastrointestinal disorders) | 23 (25) | 17 (21) | 9 (9)
Fatigue (General disorders) | 81 (99) | 40 (53) | 42 (51)
Injection Site Reaction (General disorders) | 64 (86) | 15 (16) | 26 (35)
Insomnia (General disorders) | 25 (26) | 22 (27) | 22 (24)
Allergies (Environmental or Seasonal) (Immune system disorders) | 29 (39) | 19 (21) | 18 (20)
Bronchitis (Immune system disorders) | 44 (54) | 14 (17) | 22 (30)
Cold (Immune system disorders) | 197 (358) | 102 (172) | 98 (172)
Cough (Immune system disorders) | 21 (24) | 17 (18) | 12 (13)
Flu/Flu Like Symptoms (Immune system disorders) | 98 (122) | 51 (62) | 44 (52)
GI Virus (Immune system disorders) | 33 (35) | 21 (24) | 30 (32)
Infection (General disorders) | 139 (213) | 69 (101) | 75 (122)
Sinusitis (General disorders) | 79 (120) | 32 (44) | 46 (68)
Sore Throat (General disorders) | 34 (39) | 14 (14) | 19 (22)
URI (General disorders) | 99 (148) | 53 (86) | 51 (84)
UTI (General disorders) | 64 (106) | 37 (64) | 37 (56)
Fall (Injury, poisoning and procedural complications) | 46 (63) | 20 (27) | 25 (46)
Back Pain (Musculoskeletal and connective tissue disorders) | 47 (58) | 36 (37) | 32 (40)
Joint Pain/Stiffness (Musculoskeletal and connective tissue disorders) | 40 (44) | 20 (25) | 27 (29)
Cognitive Difficulties (Nervous system disorders) | 26 (33) | 5 (5) | 18 (21)
Dizziness (Nervous system disorders) | 37 (43) | 20 (21) | 17 (22)
Extremity Pain/Soreness/Stiffness (Nervous system disorders) | 81 (105) | 41 (61) | 51 (68)
Extremity Weakness (Nervous system disorders) | 26 (34) | 10 (16) | 18 (22)
Headaches (Nervous system disorders) | 88 (116) | 40 (50) | 47 (65)
Paresthesias (Nervous system disorders) | 39 (46) | 28 (42) | 18 (18)
Unspecified Neuropathic Symptoms (Nervous system disorders) | 103 (146) | 58 (92) | 45 (67)
Anxiety/Panic Attacks (Psychiatric disorders) | 41 (48) | 20 (23) | 22 (24)
Depression (Psychiatric disorders) | 88 (103) | 40 (50) | 43 (51)
Urinary/Bladder Issues (Renal and urinary disorders) | 44 (57) | 27 (30) | 22 (25)
Dental Abcess/Extraction/Procedure (Skin and subcutaneous tissue disorders) | 43 (53) | 18 (24) | 33 (40)
Rash (Skin and subcutaneous tissue disorders) | 57 (74) | 20 (22) | 22 (25)

LIMITATIONS AND CAVEATS:
absence of a comparative randomized placebo only group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes